CLINICAL TRIAL: NCT06394570
Title: Stereotactic Treatment With neoAdjuvant Radiotherapy and Enfortumab Vedotin: a Phase I/II Study With Safety Lead-In for Localized, Cisplatin Ineligible, Muscle Invasive Bladder Cancer (STAR-EV)
Brief Title: Enfortumab Vedotin and Stereotactic Radiation for Localized, Cisplatin Ineligible Muscle Invasive Bladder Cancer
Acronym: STAR-EV
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Tian Zhang, Associate Professor- Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-0374
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — enfortumab vedotin

STUDY DESIGN:
Intervention Model Description: Safety lead-in which will assess safety of study therapy in a rule-based "escalation" approach, using the classic "3+3" design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level 0 (Experimental): Neoadjuvant therapy of Enfortumab Vedotin 1.25 mg/kg (3 cycles) and sequential Radiation Therapy starting on Cycle 3 Day 21 of EV treatment (32.5 Gray in 5 fractions)
  Interventions: Drug: Enfortumab vedotin
- Dose Level 1 (Experimental): Neoadjuvant therapy of Enfortumab Vedotin 1.25 mg/kg (3 cycles) and concurrent Radiation Therapy starting on Cycle 2 Day 15 of EV treatment (32.5 Gray in 5 fractions)
  Interventions: Drug: Enfortumab vedotin
- Dose Level 2 (Experimental): Neoadjuvant therapy of Enfortumab Vedotin 1.25 mg/kg (3 cycles) and concurrent Radiation Therapy starting on Cycle 1 Day 15 of EV treatment (32.5 Gray in 5 fractions)
  Interventions: Drug: Enfortumab vedotin

INTERVENTIONS:
Drug: Enfortumab vedotin — Enfortumab Vedotin administered 1.25mg/kg (max 125mg) IV on Day 1 and Day 8 of each 21 day cycle x 3 cycles
  Other Names: PADCEV

SUMMARY:
STAR-EV will evaluate the combination of enfortumab vedotin plus radiotherapy (RT) as neoadjuvant treatment for muscle invasive bladder cancer prior to radical cystectomy surgery. The study will use "dose escalation" to evaluate the safety and efficacy of study treatment at three dose regimens:

Level 0: EV treatment followed by RT to the bladder Level 1: EV treatment with RT starting on Cycle 2, Day 15 Level 2: EV treatment with RT starting on Cycle 1, Day 15

Following completion of EV+RT neoadjuvant therapy, all subjects will undergo surgery as part of routine care.

DETAILED DESCRIPTION:
STAR EV is a phase I/II trial with safety lead in, designed to assess safety and preliminary efficacy signal in improving pathologic complete response by adding stereotactic radiation to neoadjuvant enfortumab vedotin. Participants will be adult patients with urothelial predominant bladder cancer ineligible for neoadjuvant cisplatin-based therapy (based on provider assessment) and planned for radical cystectomy.

All participants will undergo the same treatment:

* Enfortumab vedotin (PADCEV) 1.25mg/kg (max 125mg) IV Day 1, 8 q21 day cycle x 3 cycles
* Radiation: Stereotactic radiotherapy to bladder (partial bladder volume preferred) 5 fractions; either sequential to EV treatment or concurrent with EV treatment
* Surgery: Standard of care radical cystectomy and pelvic lymph node dissection with urinary diversion per surgeon discretion.

The study will use a patient safety lead-in incorporating escalation of EV-RT from sequential to concurrent use with pre-defined stopping rules according to treatment-related adverse event (TRAE) rate of grade 3 or above. Primary endpoints are related to safety (maximum tolerated dose "regimen" based on dose limiting toxicities (DLTs) observed) and pathologic complete response rate at the time of surgery. Subjects will be followed for one year following cystectomy, or completion of neoadjuvant therapy for any subject who does not undergo cystectomy for any reason.

ELIGIBILITY:
Inclusion Criteria:

1. Urothelial carcinoma of the urinary bladder stage cT2-4a (AJCC 8th edition) N0M0 planned for radical cystectomy. Mixed cell types with variant histologies (including squamous, plasmacytoid, adenocarcinoma, sarcomatoid, micropapillary, nested, and lipid cell variants) are allowed as long as any urothelial histology is present (i.e. -not 100% variant histology). Small cell/neuroendocrine component is excluded.
2. Ineligibility for cisplatin-based chemotherapy based on treating physician assessment and any of the following "Galsky criteria": renal insufficiency (Creatinine Clearance <60ml/min by standard institutional calculation method), >=grade 2 peripheral neuropathy, >=grade 2 hearing loss, New York Heart Association (NYHA) class III heart failure; a combination of these; or patient refusal.
3. Age >=18.
4. Performance status Eastern Cooperative Oncology Group (ECOG) 0-1
5. Adequate organ and marrow function as defined below:

   •Hematologic:

   -Absolute neutrophil count (ANC) >=1500/mm3
   * Platelet count >=100x109/L
   * Hemoglobin ≥ 9 g/dL

     •Hepatic:
   * Serum bilirubin ≤ 1.5 × upper limit of normal (ULN) or ≤ 3 × ULN for subjects with Gilbert's disease
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN

     •Renal:
   * No end stage renal disease requiring dialysis allowed
6. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 3 months following completion of study neoadjuvant therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

6a. A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

  7.Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. No prior systemic therapy (except prior therapy for non-muscle invasive bladder cancer >12 prior to registration) for bladder cancer or prior pelvic radiotherapy. Prior intra-vesical therapies are allowed, including Bacillus Calmette-Guerin (BCG) for non-muscle invasive bladder cancer. Prior chemotherapy for other cancers is allowed if given >=1 year prior to study registration.
2. Baseline >= Grade 2 sensory or motor neuropathy
3. Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to enfortumab vedotin or other agents used in study.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
6. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) Regimen | From initiation of Enfortuman Vedotin treatment until post neoadjuvant therapy visit (approximately 120 days)
  A standard 3 + 3 dose escalation schedule will be used for all escalations. Enfortumab Vedotin will be given for three 21 day cycles. Radiation therapy will be administered at dose level 0, level 1 or level 2.
Pathologic Complete response rate at radical cystectomy | At radical cystectomy following completion of neoadjuvant therapy (approximately 6 weeks after completion of EV treatment)
  Rate of complete pathologic response in bladder tumor biopsy at cystectomy according to postsurgical staging.

SECONDARY OUTCOMES:
Adverse Events | From initiation of neoadjuvant therapy to completion of final post treatment study visit (approximately 4 months)
  Adverse events reported and observed according to CTCAE v5.0
Rate of pathologic downstaging in the bladder | At radical cystectomy following completion of neoadjuvant therapy (approximately 6 weeks after completion of EV treatment)
  Rate of post surgical pathologic staging being less than clinical staging.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided